CLINICAL TRIAL: NCT06090578
Title: A Pragmatic Trial of the TabCAT Brain Health Assessment for the Detection of Cognitive Impairment in Primary Care
Brief Title: TabCAT Brain Health Assessment in Primary Care
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Kaiser Permanente (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: U01NS128913 (NIH); U01NS128913 (NIH)
Record Dates: First submitted 2023-10-13; First posted 2023-10-19 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Mild Cognitive Impairment; Dementia
Keywords: Primary care; Cognitive assessment
MeSH Terms: conditions — Cognitive Dysfunction; Dementia

STUDY DESIGN:
Intervention Model Description: This is a pragmatic cluster randomized trial. 26 primary care clinics will be randomized in two 18-month waves to receive either the TabCAT-BHA paradigm or usual care. The first wave will include six intervention practices and the second wave will include seven intervention practices.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TabCAT-Brain Health Assessment Clinical Pathway (Experimental): Primary care providers concerned that their patients are exhibiting signs of cognitive decline based on patient, informant (family), or provider concerns will refer them for a TabCAT-BHA assessment and follow-up care.
  Interventions: Other: TabCAT Brain Health Assessment Clinical Pathway
- Usual Care Clinical Pathway (No Intervention): Patients in the control practices will continue with usual care workflows.

INTERVENTIONS:
Other: TabCAT Brain Health Assessment Clinical Pathway — Primary care providers concerned that their patients are exhibiting signs of cognitive decline will refer them to clinical associates who will then perform the TabCAT-BHA tablet-based test. The TabCAT-BHA paradigm comprises 7-10 minutes of tablet-based testing and an optional 3-minute self-administered informant survey captures behavioral symptoms and change from baseline. The results are available to the PCP in the EMR along with turnkey guidance to evaluate for reversible causes, identify and involve a care partner, make and disclose diagnosis, provide community and educational resources, and make medical referrals as appropriate. Nursing support is available to support the PCP in making the diagnosis and to consult to the family via telephone post-diagnosis to address immediate care needs.
  Arms: TabCAT-Brain Health Assessment Clinical Pathway

SUMMARY:
Efficient and user-friendly paradigms to detect cognitive impairment, including dementia are needed in primary care. The TabCAT Brain Health Assessment accurately detects cognitive impairment via an appealing tablet interface with automated scoring and EMR integration. This study will evaluate the effectiveness of the paradigm on detection rates and other brain health outcomes via a pragmatic cluster randomized trial in 26 Kaiser Southern California primary care clinics.

DETAILED DESCRIPTION:
Twenty-six Kaiser Permanente Southern California (KPSC) primary care clinics will be randomized in two waves to receive either the TabCAT-BHA paradigm or usual care. Clinics have been matched in pairs by number of providers, median panel size, the racial/ethnic makeup of the patient panel, baseline rates of cognitive impairment diagnosis, rates of telehealth encounters, and percentage of members who are 65+ in the practice. The trial will be conducted over two 18-month waves, with six intervention practices in the first wave and seven intervention practices starting in the second wave. All patients seen at least once across these 26 practices will be included in the trial and the primary analyses will use data extracted from the EMR. Patients in the intervention practices will receive care in accordance with the TabCAT-BHA paradigm whereas patients in the control practices will continue with usual care workflows. The intervention will include a 6-month startup period during which the research team will partner with the physician leads to adapt the paradigm workflows to each practice and onboard the PCPs, and then a 12-month steady state period when effectiveness on the primary and secondary outcomes will be measured. During the TabCAT-BHA paradigm intervention, pragmatically, primary care providers concerned that their patients are exhibiting signs of cognitive decline will refer them to clinical research associates located in the primary care clinics who will then perform the TabCAT-BHA tablet-based test either on the spot or as a scheduled procedure visit. The tablet-based test provides an automated scoring report that includes guidance for providers to identify reversible causes of cognitive impairment, involving a care partner, diagnostic disclosure, community and educational resources, and specialty referral including the option to refer the patient for a "Brain Health Consultation" telephone call with a study nurse or social worker.

ELIGIBILITY:
Inclusion Criteria:

* Patient with at least one encounter at an intervention clinic during the intervention period
* Age 18+ (limited to 65+ for primary analyses)

Exclusion Criteria:

* Patients under the age of 18.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180000 (Estimated)
Dates: Start 2023-07-27 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The rate of patients with at least one cognitive impairment diagnosis documented in the medical record by any primary care provider during the 12-month steady state period at the clinic. | During the 12-month steady state period
  Rate is out of all patients with an encounter during the steady state period at the clinic. The primary analyses for all outcomes are limited to ages 65+.

SECONDARY OUTCOMES:
The rate of patients who have a documented standardized cognitive assessment performed in the primary care clinic within 4 months of an incident cognitive impairment diagnosis. | During the 12-month steady state period
  Rate is out of all patients with an encounter at the clinic during the 12-month steady state period and an incident cognitive impairment diagnosis. The window for incident cognitive impairment diagnoses will be the steady state period + 4 months after. The standardized cognitive assessment must occur during the steady state period and +/- 4 months of the incident diagnosis. All standardized cognitive assessments will be counted. Incident diagnoses are the first time that any of these diagnoses are documented in the medical record by any outpatient provider, using a 2 year look back window. In addition, incident diagnoses of mild cognitive impairment and dementia will be counted even if an "other cognitive impairment diagnosis" was previously made.
The rate of patients who have a referral to Geriatrics, Neurology or Psychiatry. | During the 12-month steady state period
  Rate is out of all patients with an incident diagnosis, as defined in Outcome 2. The referral must occur within the 12-month steady state period + 4 months after, and within +/- 4 months of the incident diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Possin, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- Kaiser Permanente Southern California Department of Research & Evaluation, Pasadena, California, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared outside of Kaiser Permanente Southern California.

REFERENCES:
- [Result] Bernstein Sideman A, Chalmer R, Ayers E, Gershon R, Verghese J, Wolf M, Ansari A, Arvanitis M, Bui N, Chen P, Chodos A, Corriveau R, Curtis L, Ehrlich AR, Tomaszewski Farias SE, Goode C, Hill-Sakurai L, Nowinski CJ, Premkumar M, Rankin KP, Ritchie CS, Tsoy E, Weiss E, Possin KL. Lessons from Detecting Cognitive Impairment Including Dementia (DetectCID) in Primary Care. J Alzheimers Dis. 2022;86(2):655-665. doi: 10.3233/JAD-215106. PMID 35124639
- [Derived] Sideman AB, Nguyen HQ, Langer-Gould A, Lee EA, Borson S, Shen E, Tsoy E, Macias M, Goode C, Rankin K, Kramer J, Possin KL. Stakeholder-informed pragmatic trial protocol of the TabCAT-BHA for the detection of cognitive impairment in primary care. BMC Prim Care. 2024 Aug 6;25(1):286. doi: 10.1186/s12875-024-02544-9. PMID 39107706